CLINICAL TRIAL: NCT04466540
Title: Pragmatic, Double-blind, Placebo-controlled Randomized Clinical Trial, Evaluating Hydroxychloroquine for Prevention of Hospitalization and Respiratory Complications in Non-hospitalized Patients With Confirmed or Probable COVID-19
Brief Title: Randomized Placebo-controlled Trial of Hydroxychloroquine in Outpatient Cases With Coronavirus Disease 2019 (COVID-19)
Acronym: COALITION-V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Collaborators: EMS S/A (Unknown); Hospital do Coracao (Other); Hospital Israelita Albert Einstein (Other); Hospital Sirio-Libanes (Other); Hospital Moinhos de Vento (Other); Brazilian Research In Intensive Care Network (Network)
Responsible Party: Principal Investigator, Álvaro Avezum Junior, Research Manager - International Research Center, Hospital Alemão Oswaldo Cruz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30415320.8.1001.0070
Record Dates: First submitted 2020-07-03; First posted 2020-07-10 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: COVID-19; Severe Acute Respiratory Syndrome - Coronavirus-2; Hydroxychloroquine; COALITION Brazil V 2019; Outpatients
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Pragmatic, double-blind, placebo-controlled randomized parallel-group, two-arm clinical trial (with allocation ratio 1:1)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization (1:1) is generated by a validated software and performed in permuted blocks of size 8. Concealment of the randomization list is maintained through a 24-hour, centralized, automated, internet-based randomization system. Furthermore, as placebo-controlled study, the placebo will have the same structural characteristics as the active drug and will be dispensed in cartridges that do not allow the identification of what is being given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (HCQ) (Experimental): HCQ group participants will receive a dose of 400mg twice daily (BID) in the first day, and a dose of 400 mg once daily (OD) from the second day of treatment, in a total of 7 days.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): The placebo group will follow the same regimen of administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine pharmaceutical form will be tablets of 400 mg.
  Arms: Hydroxychloroquine (HCQ)
Drug: Placebo — Hydroxychloroquine placebo
  Arms: Placebo

SUMMARY:
In December 2019, a group of patients with pneumonia of unknown cause was identified in Wuhan, in the Hubei province, China. Despite the need of target specific therapeutic options for COVID-19, until now there is no proof of effectiveness of any specific intervention. Some limited observational trials and also evidence from randomized trials have shown no benefit of hydroxychloroquine in inpatient context. Thus, studies evaluating interventions in an outpatient setting in non-severe patients can provide important information related to prognosis and safety. In this way, the present study will evaluate the effectiveness and safety of the use of hydroxychloroquine in COVID-19 outpatients by means of a Randomized, double-blind, placebo-controlled trial

DETAILED DESCRIPTION:
Pragmatic, double-blind, placebo-controlled randomized parallel-group, two-arm clinical trial (with allocation ratio 1:1), evaluating hydroxychloroquine (800 mg at 1st day, and 400 mg from day 2 to 7) for prevention of hospitalization and respiratory complications in non-hospitalized confirmed or suspected COVID-19 cases. Key inclusion criteria are adults (equal to or greater tahn 18 years) seeking medical care with suspected or confirmed COVID-19, with time between symptoms and inclusion ≤ 07 days, presenting mild symptoms, without indication of hospitalization and at least one risk factor for complication (> 65 years; hypertension; diabetes mellitus; asthma; Chronic Obstructive Pulmonary Disease (COPD) or other chronic lung diseases; smoking; immunosuppression; obesity (Defined as BMI equal to or greater than 30 Kg/m2). Primary endpoint is to assess if the treatment with hydroxychloroquine is able to avoid hospitalization due to a COVID-19-related clinical reason within 30 days of randomization in an outpatient setting. Hospitalization is considered to be hospital stay for a period > 24h or an additional hospitalized calendar day. The primary endpoint is centrally adjudicated by an independent clinical events committee blinded to the assigned treatment groups. Secondary endpoints include uncontrolled asthma after ≥ 5 days of starting study medication; pneumonia; otitis media; fever resolution time; time to improve respiratory symptoms; hospitalization in the Intensive Care Unit; need for orotracheal intubation; mechanical ventilation time; mortality. Safety outcomes will be hypoglycemia; palpitations; reduced visual acuity; diarrhea; anorexia; and emotional lability. The evaluation of the primary outcome (hospitalization within 30 days) will be performed for the included population following the principle of intention-to-treat (ITT), which will consist of all randomized cases. A modified intention-to-treat analysis (mITT), in which cases definitely confirmed as negative for COVID-19 will be excluded, will also be performed.

ELIGIBILITY:
Inclusion Criteria:

It will be considered eligible those adults (equal to or greater than 18 years) seeking medical care with suspected or confirmed COVID-19, with time between symptoms and inclusion ≤ 07 days, presenting mild symptoms, without indication of hospitalization and at least 1 risk factor for complication:

1. > 65 years;
2. Hypertension;
3. Diabetes mellitus;
4. Asthma;
5. COPD or other chronic lung diseases;
6. Smoking;
7. Immunosuppression;
8. Obesity (Defined as BMI equal to or greater than 30 Kg/m2).

Exclusion Criteria:

1. Patients under 18 years old;
2. Hospitalization at the first medical care;
3. Positive test for influenza at the first medical care;
4. Known hypersensitivity to hydroxychloroquine / chloroquine;
5. Previous diagnosis of retinopathy or macular degeneration;
6. Previous diagnosis of Long QT-syndrome, history of sudden death in close family members (parents and siblings), decompensated heart failure, unstable coronary artery disease, use of anti-arrhythmic drugs or other drugs that can increase the hydroxychloroquine bioavailability or enhance its effect;
7. Evidence of known liver disease, reported by the patient;
8. Evidence of known chronic kidney disease, reported by the patient;
9. Patients with pancreatitis;
10. Baseline ECG with QTc interval ≥ 480ms;
11. Chronic use of hydroxychloroquine/chloroquine for other reasons;
12. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Hospitalization | 30 days from randomization
  To assess if the treatment is able to avoid hospitalization due to a COVID-19-related clinical reason within 30 days of randomization in an outpatient setting. Hospitalization is considered to be hospital stay for a period > 24h or an additional hospitalized calendar day.

SECONDARY OUTCOMES:
Uncontrolled asthma after ≥ 5 days of starting study medication | within 30 days from randomization
  Affirmative answer in three or four items of the Global Initiative for Asthma (GINA) questionnaire
Pneumonia | within 30 days from randomization
  Defined by clinical-radiological criteria - a history of cough and one or more of the following symptoms: sputum, dyspnea, chest pain, sweating or fever (T> 37.8o C) + Chest CT scan showing ground-glass opacity, focal consolidations or mixed opacities (including reverse halo sign), uni or bilateral
Otitis media | within 30 days from randomization
  Defined by clinical criteria - Fever (T> 37.8o C) and otalgia + bulging of the tympanic membrane
Fever resolution time | within 30 days from randomization
  Day 0 of fever resolution will be defined as the first afebrile day (T <37.5o C) after inclusion in the study followed by at least two consecutive days. The temperature will be obtained through the participant report in the patient's diary
Time to improve respiratory symptoms | within 30 days from randomization
  Time to improve respiratory symptoms (cough, runny nose)
Hospitalization in the Intensive Care Unit | within 30 days from randomization
  Admission to ICU due to clinical reasons related to COVID-19
Need for Orotracheal Intubation | within 30 days from randomization
  Clinical need for Orotracheal Intubation as assessed by the physician responsible for the case
Mechanical Ventilation Time | within 30 days from randomization
  Number of days on mechanical ventilation until extubation or death
Mortality | within 30 days from randomization
  Death due to any cause that occurred within 30 days after inclusion in the study

OTHER OUTCOMES:
Hypoglycemia | within 30 days from randomization
  Change in the frequency of hypoglycemic episodes in diabetic patients using hypoglycemic medication, perceived by clinical signs or symptoms or measured in a capillary or blood glucose device
Palpitations | within 30 days from randomization
  Presence of cardiac arrhythmias in patients without known history of prolongation of the measure between Q wave and T wave in the heart's electrical cycle (QTc) or pre-existing heart disease;
Reduced visual acuity | within 30 days from randomization
  Change in visual acuity or new diagnosis of retinal disease not previously documented
Diarrhea | within 30 days from randomization
  Change in bowel habit greater than three (3) diarrheal episodes per day during the use of hydroxychloroquine medication and 3 days after its end
Anorexia | within 30 days from randomization
  Change in appetite during medication use hydroxychloroquine and 3 days after the end of treatment
Emotional lability | within 30 days from randomization
  Perception of change in emotional lability (mood swings) during hydroxychloroquine use and 3 days after the end of treatment
Time to hospitalization after randomization | within 30 days from randomization
  Time from randomization to hospitalization
Assessment of the patient clinical status at the time of hospitalization | within 30 days from randomization
  Clinical and vital signs assessed when admitted to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Avezum, Ph.D, Principal Investigator — International Research Center - Hospital Alemão Oswaldo Cruz
Locations (69):
- Brazil (69):
  - Centro de Pesquisas Clínicas Dr. Marco Mota HCOR, Maceió, Alagoas
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Hospital Unimed Cariri, Juazeiro do Norte, Ceará
  - Unimed Sul Capixaba, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital e Clínica São Roque, Ipiaú, Estado de Bahia
  - Clínica Otorhinus, Salvador, Estado de Bahia
  - Hospital da Bahia, Salvador, Estado de Bahia
  - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Instituto Cárdio Pulmonar da Bahia, Salvador, Estado de Bahia
  - Hospital SAMUR, Vitória da Conquista, Estado de Bahia
  - Hospital das Clínicas Universidade Federal de Goiás, Goiânia, Goiás
  - Santa Casa de Misericórdia de Passos, Passos, Minas Agerais
  - Hospital Júlia Kubitschek, Belo Horizonte, Minas Gerais
  - Instituto da Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Casa de Caridade de Carangola, Carangola, Minas Gerais
  - Hospital Maternidade e Pronto Socorro Santa Lucia, Poços de Caldas, Minas Gerais
  - Hospital da Unimed, São João del Rei, Minas Gerais
  - Santa Casa de Misericórdia de São João Del Rei, São João del Rei, Minas Gerais
  - Hospital de Clínicas da Universidade Federal do Triangulo Mineiro, Uberaba, Minas Gerais
  - Hospital de Clínicas da Universidade Federal de Uberlândia, Uberlândia, Minas Gerais
  - Hospital do Rocio, Campo Largo, Paraná
  - Clínica Clinilive, Maringá, Paraná
  - Hospital Universitário Regional de Maringá, Maringá, Paraná
  - PROCAPE, Recife, Pernambuco
  - Real Hospital Português de Beneficência em Pernambuco, Recife, Pernambuco
  - SECRETARIA MUNICIPAL DE SAÚDE DE SAIRÉ (Unidade Mista Olília Mendonça Souto Maior), Sairé, Pernambuco
  - Complexo Hospitalar de Niterói, Niterói, Rio de Janeiro
  - Hospital Unimed Volta Redonda, Volta Redonda, Rio de Janeiro
  - Associação Dr. Bartholomeu Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Misericórdia de Porto Alegre (ISCMPA), Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Santa Maria, Santa Maria, Rio Grande do Sul
  - CEPEM Centro de Pesquisa de Medicina Tropical de Rondônia, Porto Velho, Rondônia
  - Irmandade de Misericórdia Do Hospital Da Santa Casa de Monte Alto, Monte Alto, Salto Alto
  - Maestri e Kormann Consultoria Medico Cientifica, Blumenau, Santa Catarina
  - Imigrantes Hospital e Maternidade, Brusque, Santa Catarina
  - Hospital São José, Criciúma, Santa Catarina
  - Hospital Regional Hans Dieter Schmidt, Joinville, Santa Catarina
  - Santa Casa de Araras, Araras, São Paulo
  - Hospital de Amor, Barretos, São Paulo
  - Santa Casa de Misericórdia de Barretos, Barretos, São Paulo
  - Alphacor Cardiologia Clinica E Diagnóstica LTDA, Barueri, São Paulo
  - Faculdade de Medicina de Botucatu, UNESP, Botucatu, São Paulo
  - Hospital Regional do Litoral Norte, Caraguatatuba, São Paulo
  - Hospital de Cordeirópolis, Cordeirópolis, São Paulo
  - Centro de Combate ao Coronavírus de Itapevi, Itapevi, São Paulo
  - Dux Medicina, Jundiaí, São Paulo
  - Hospital Carlos Fenando Malzoni, Matão, São Paulo
  - Centro de Atendimento Para O Enfrentamento A Covid-19 Da Prefeitura Municipal de Monte Altoprefeitura de Monte Alto, Monte Alto, São Paulo
  - Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Unimed Ribeirão Preto, Ribeirão Preto, São Paulo
  - Hospital Casa de Saúde de Santos, Santos, São Paulo
  - Kaiser Clínica e Hospital Dia, São José do Rio Preto, São Paulo
  - Hospital Policlin, São José dos Campos, São Paulo
  - Hospital Regional de São José dos Campos, São José dos Campos, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga, São Paulo
  - ESF Dr. João Paccola Primo, Lençois Paulista
  - Cardioclinica da Ilha do Governador, Rio de Janeiro
  - International Research Center - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital do Coração, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital Leforte, São Paulo
  - Hospital Moriah, São Paulo
  - Hospital Samaritano, São Paulo
  - Hospital Santa Paula, São Paulo
  - Hospital São Camilo Pompéia, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo
  - Hospital Sírio-Libanês, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avezum A, Oliveira GBF, Oliveira H, Lucchetta RC, Pereira VFA, Dabarian AL, D O Vieira R, Silva DV, Kormann APM, Tognon AP, De Gasperi R, Hernandes ME, Feitosa ADM, Piscopo A, Souza AS, Miguel CH, Nogueira VO, Minelli C, Magalhaes CC, Morejon KML, Bicudo LS, Souza GEC, Gomes MAM, Fo JJFR, Schwarzbold AV, Zilli A, Amazonas RB, Moreira FR, Alves LBO, Assis SRL, Neves PDMM, Matuoka JY, Boszczowski I, Catarino DGM, Veiga VC, Azevedo LCP, Rosa RG, Lopes RD, Cavalcanti AB, Berwanger O; COPE - COALITION COVID-19 Brazil V Investigators. Hydroxychloroquine versus placebo in the treatment of non-hospitalised patients with COVID-19 (COPE - Coalition V): A double-blind, multicentre, randomised, controlled trial. Lancet Reg Health Am. 2022 Jul;11:100243. doi: 10.1016/j.lana.2022.100243. Epub 2022 Mar 31. PMID 35378952
- [Derived] Oliveira Junior HA, Ferri CP, Boszczowski I, Oliveira GBF, Cavalcanti AB, Rosa RG, Lopes RD, Azevedo LCP, Veiga VC, Berwanger O, Avezum A. Rationale and Design of the COVID-19 Outpatient Prevention Evaluation (COPE - Coalition V) Randomized Clinical Trial: Hydroxychloroquine vs. Placebo in Non-Hospitalized Patients. Arq Bras Cardiol. 2022 Feb;118(2):378-387. doi: 10.36660/abc.20210832. English, Portuguese. PMID 35262569